CLINICAL TRIAL: NCT05547178
Title: Self-perceived Changes in Everyday Life Among Participants of a Fall Prevention Study With Tai Chi or Eurythmy Intervention Versus Standard Care: a Qualitative Exploration as a Sub-Study of the ENTAiER Study
Brief Title: Changes in Everyday Life After a Tai Chi or Eurythmy Intervention in Elderly People at Risk of Falling: a Qualitative Exploration as a Sub-Study of the ENTAiER Study
Status: Completed | Type: Observational
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: EYT_13
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Increased Risk of Falls
Keywords: Old age; Chronic disease; Risk of falls; Fear of falling; Fall prevention; Eurythmy; Tai Chi
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Eurythmy Therapy (performed as part of the ENTAiER main study)
  Interventions: Other: Qualitative interview - eurythmy group
- Tai Chi (performed as part of the ENTAiER main study)
  Interventions: Other: Qualitative interview - tai chi group
- Standard Care
  Interventions: Other: Qualitative interview - standard care group

INTERVENTIONS:
Other: Qualitative interview - eurythmy group — Participants will be interviewed about self-perceived changes in everyday life during participation in the eurythmy intervention of the ENTAiER study.
  Groups: Eurythmy Therapy (performed as part of the ENTAiER main study)
Other: Qualitative interview - tai chi group — Participants will be interviewed about self-perceived changes in everyday life during participation in the tai chi intervention of the ENTAiER study.
  Groups: Tai Chi (performed as part of the ENTAiER main study)
Other: Qualitative interview - standard care group — Participants will be interviewed about self-perceived changes in everyday life during participation in the standard care group of the ENTAiER study.
  Groups: Standard Care

SUMMARY:
The ENTAiER fall prevention study investigates the efficacy and safety of eurythmy therapy and tai chi in older people with chronic diseases and an increased risk of falls. In the course of the ENTAiER study, the participants observed changes in themselves and in their everyday life and described them in conversation, which could not be recorded with the research methods used. A qualitative exploration of these subjectively experienced changes among participants of the ENTAiER study will be conducted as part of a sub-study. For this purpose, group interviews will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled and randomized participant of ENTAiER main study
* Written informed consent for participation in EYT_13 sub-study
* Participation in eurythmy or tai chi intervention for 24 weeks (-28d/+21d) (the standard care group will be time-equated to eurythmy and tai chi)

Exclusion Criteria:

* Early termination of the intervention (less than 20 weeks) (the standard care group will be time-equated to eurythmy and tai chi)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects who have consented to participate and are enrolled in the ENTAiER main study will be approached for participation in this sub-study. Sub-study will be conducted at the ARCIM Institute, Filderstadt.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Self-reported changes in daily life through movement exercises | 90-minute interviews
  Semi-structured guided group interviews will be used

SECONDARY OUTCOMES:
Self-reported changes in the experience of movement in general | 90-minute interviews
  Semi-structured guided group interviews will be used
Self-reported changes in movement security through movement exercises | 90-minute interviews
  Semi-structured guided group interviews will be used
Self-reported changes in health through movement exercises | 90-minute interviews
  Semi-structured guided group interviews will be used
Integration of movement exercises into everyday life | 90-minute interviews
  Semi-structured guided group interviews will be used
Experiencing movement exercises | 90-minute interviews
  Semi-structured guided group interviews will be used
Need for offers on movement exercises | 90-minute interviews
  Semi-structured guided group interviews will be used

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr, Principal Investigator — ARCIM Institute
Locations (1):
- Arcim Institute, Filderstadt, Baden-Wurttemberg, Germany